CLINICAL TRIAL: NCT04049162
Title: Effects of Blueberry Consumption on Vascular Function, Physical Activity, and Cognition in Sedentary Older Adults
Brief Title: Blueberry Enhances Activity and Cognition Through Increased Vascular Efficiency
Acronym: BEACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00101714
Record Dates: First submitted 2019-07-23; First posted 2019-08-08 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Sedentary Lifestyle; Blood Pressure; Arterial Stiffness; Overweight and Obesity
Keywords: Blueberries; Pulse Wave Velocity; Aging; Exercise; Cognition
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity; Motor Activity | interventions — blueberry extract; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry Plus Exercise (BB-EX) (Experimental): BB-Ex participants will consume lyophilized blueberry powder, mixed with water (18 grams, equivalent to 3/4ths cup of blueberries) with 2 daily meals (36 g/d blueberry powder total; approx. 1.5 servings/d)
  Interventions: Dietary Supplement: Blueberry Plus Exercise (BB-EX)
- Blueberry Placebo Plus Exercise (P-EX) (Placebo Comparator): Participants randomized to P-EX treatment will consume an indistinguishable placebo powder, matched for color, flavor, consistency, and caloric content, in the same manner.
  Interventions: Dietary Supplement: Blueberry Placebo Plus Exercise (P-EX)

INTERVENTIONS:
Dietary Supplement: Blueberry Plus Exercise (BB-EX) — Pre-packaged blueberry powders are from U.S. Highbush Blueberry Council and are packaged in sealed single-serving packets (18 g/packet) to prevent exposure to light and moisture. All supplement packets are stored under refrigeration until distribution to study participants. Participants will be asked to increase physical activity through a weekly supervised exercise class and increasing baseline daily step counts gradually over the course of the intervention.
  Other Names: Lyophilized Blueberry Powder
  Arms: Blueberry Plus Exercise (BB-EX)
Dietary Supplement: Blueberry Placebo Plus Exercise (P-EX) — Pre-packaged placebo powders are from U.S. Highbush Blueberry Council and are packaged in sealed single-serving packets (18 g/packet) to prevent exposure to light and moisture. All supplement packets are stored under refrigeration until distribution to study participants. Participants will be asked to increase physical activity through a weekly supervised exercise class and increasing baseline daily step counts gradually over the course of the intervention.
  Other Names: Placebo Blueberry Powder
  Arms: Blueberry Placebo Plus Exercise (P-EX)

SUMMARY:
Recent evidence suggests that increased berry intake results in a variety of health benefits, across multiple health domains. This 3-month randomized, double-blind, placebo-controlled trial assess the effects of combining daily blueberry intake with weekly exercise (BB-EX) on cardiovascular function, as well as physical activity and cognitive function, in sedentary older adults (>60 years). We will compare these effects to the same outcomes with a control group consuming a blueberry placebo (P-EX) at 0, 4, 8 and 12 weeks.

DETAILED DESCRIPTION:
A 12-week randomized, double-blind, placebo-controlled physical activity intervention will be administered in sedentary older (>60 years) women and men randomized to either lyophilized blueberry powder, rehydrated and consumed as a beverage twice daily with meals (BB-EX; n = 25), or an indistinguishable placebo powder, taken in the same manner (placebo control; P-EX; n = 25).

Vascular function (primary outcome), 24-hr ambulatory blood pressure, cognitive performance, and related secondary measures will be assessed at 0 and 12 weeks; berry and nutrient intake and function are assessed every 4 weeks; and physical activity as step counts will be continuously monitored using a mobile device (Garmin). Blood, urine (24-hr), and stool samples will be collected at 0 and 12 weeks and archived for later analysis.

The 12-week study duration is based upon the timing of vascular responses seen in other trials, as well as the minimal time needed to expect a change in cognitive performance in an older adult population. The blueberry dose of 36 grams per day in a split dose consumed with meals is based on (1) a 33% increase in dose over that previously used in a longer (6-month) trial; (2) delivering the most effective dose of blueberry bioactives; and (3) reduced likelihood of any gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Overweight (BMI ≥25 to 35 kg/m2)
* Well-controlled blood pressure (< 150/90 mmHg)
* Able to speak and understand spoken and written English
* Cognitively normal (Mini-Cog score 3-5)
* Able to walk independently
* Social security number (required for compensation)
* Own a smartphone or other mobile device capable of downloading the Garmin Connect app

Exclusion Criteria:

* Exercise > 150 minutes/week
* Unwillingness or inability to be randomized to any one of two intervention groups without knowing which (double-blind), submit to all study testing, or continuously participate in a randomly assigned diet and exercise intervention for six months.
* Unwilling to restrict consumption of anthocyanin-rich foods
* Unwillingness to abstain from mood altering drugs (including marijuana but excluding CBDs) for 7 days prior to baseline and endpoint testing.
* Self-reported vegetarian or vegan.
* Inability to complete written recording forms including journals of eating and exercise behaviors.
* Inability to complete written and computerized cognitive tasks (presented in English).
* Allergy or intolerance to blueberry or placebo powder ingredients Placebo ingredients include: maltodextrin, fructose, artificial blueberry flavor, natural blueberry flavor, artificial purple color (water, FD&C Red #40, FD&C Blue #1, malic acid, sodium benzoate) citric acid, and artificial red color (water, FD&C Red #40, malic acid, sodium benzoate, silica dioxide).
* Gastrointestinal disorders that influence digestion and absorption of food, e.g., IBD
* History of frequent urinary tract or Clostridium difficile infections
* Presence of unstable, acutely symptomatic, or life-limiting illness.
* Regular use of medication that interferes with the measurement of study outcomes as determined by the study physician.
* Unstable use of medications, other than statins, for conditions associated with metabolic syndrome (hypertension, diabetes, dyslipidemia) during the prior 6 months or during the study.
* Antibiotic use in the last 3 months.
* Cigarette smoking, chewing, or use of nicotine replacement products in the past 3 months or during the course of the study.
* Colonoscopy in last 2 months.
* History of stomach or bowel resection (other than appendectomy), gastric bypass or other bariatric weight loss procedure effecting absorption.
* History of significant weight instability (defined as > 10 pounds weight gain or loss over one month prior to study participation).
* History of cancer treatment (other than melanoma skin cancer) and not "cancer-free" for at least 1 year.
* History of anti-hormonal therapy (eg., for breast or prostate cancer) within the last 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pulse wave velocity at 12 weeks | 0 to 12 weeks
  Change in carotid-femoral pulse wave velocity will be assessed using applanation tonometry, (SphygmoCor Pulse Wave Velocity System)

SECONDARY OUTCOMES:
Change from baseline in cognitive flexibility at 12 weeks | 0 to 12 weeks
  Change in cognitive performance will be assessed using a computerized task-switching test in which participants predictably alternate between two discrimination tasks.
Change from baseline in physical activity at 12 weeks | 0 to 12 weeks
  Change in physical activity will be measured using a commercial activity monitor, which will be worn 24 hr/d to capture total daily steps as the measure of physical activity.
Change from baseline in ambulatory blood Pressure at 12 weeks | 0 to 12 weeks
  Change in ambulatory blood pressure will be measured using an Ambulatory BP Monitor, with readings taken every 30 min. during the day and 60 min. at night, over a 24-hour period.
Change from baseline in total calories at 4, 8 and 12 weeks | 0 to 12 weeks (0, 4, 8 and 12 weeks)
  Total calories will be measured using 3-day food records (participants record everything they eat and drink for three days)
Change from baseline in macronutrient intake at 4, 8 and 12 weeks | 0 to 12 weeks (0, 4, 8 and 12 weeks)
  Total calories will be measured using 3-day food records (participants record everything they eat and drink for three days)
Change from baseline in micronutrient intake at 4, 8 and 12 weeks | 0 to 12 weeks (0, 4, 8 and 12 weeks)
  Total calories will be measured using 3-day food records (participants record everything they eat and drink for three days)
Change from baseline aerobic endurance at 4, 8, and 12 weeks | 0 to 12 weeks (0, 4, 8 and 12 weeks)
  Change in aerobic endurance will be determined by a 6-minute walk where subjects walk as many laps as possible in 6 minutes between cones placed 100 feet apart.
Change from baseline hand grip strength at 4, 8 and 12 weeks | 0 to 12 weeks (0, 4, 8 and 12 weeks)
  Change in maximal upper body strength will be determined using hydraulic isometric hand dynamometer.

OTHER OUTCOMES:
Change from baseline in central arterial pressure at 12 weeks | 0 to 12 weeks
  Change in central arterial pressure waveform will be assessed using an automated brachial cuff.
Baseline dietary intake (Total calories) | 0 weeks
  Average caloric intake will be assessed using the Diet History Questionnaire III (NCBI) food frequency questionnaire.
Baseline dietary intake (macronutrient intake) | 0 weeks
  Average Macronutrient intake will be assessed using the Diet History Questionnaire III (NCBI) food frequency questionnaire.
Baseline dietary intake (micronutrient intake) | 0 weeks
  Average micronutrient intake will be assessed using the Diet History Questionnaire III(NCBI) food frequency questionnaire.
Change from baseline in body weight | 0 to 12 weeks
  Change in body weight will be assessed weekly using the same scale, light clothing and no shoes.
Height at baseline | 0 weeks
  Height will be measured using a wall-mounted stadiometer.
Seated blood pressure at baseline | 0 weeks
  Seated systolic and diastolic blood pressure will be measured, in duplicate, using an digital blood pressure monitor following 5 minutes of quiet sitting.
Change from baseline verbal memory at 12 weeks | 0 to 12 weeks
  Verbal learning and memory will be assessed using the Hopkins Verbal Learning Test.
Change from baseline Executive Function at 12 weeks | 0 to 12 weeks
  Executive function will be assessed using the Trail Making Test.
Change from baseline processing speed at 12 weeks | 0 to 12 weeks
  Change in processing speed will be assessed using the Symbol Digit Modalities Test (SDMT).
Change from baseline reaction time at 12 weeks | 0 to 12 weeks
  Change in reaction time will be assessed by computerized test using CANTAB (www.cambridgecognition.com).
Change from baseline paired associates learning at 12 weeks | 0 to 12 weeks
  Change in paired associates learning will be assessed by computerized test using CANTAB (www.cambridgecognition.com).
Change from baseline spatial working memory at 12 weeks | 0 to 12 weeks
  Change in spatial working memory will be assessed by computerized test using CANTAB (www.cambridgecognition.com).
Change from baseline pattern recognition memory at 12 weeks | 0 to 12 weeks
  Change in pattern recognition memory will be assessed by computerized test using CANTAB (www.cambridgecognition.com).
Change from baseline delayed matching to sample at 12 weeks | 0 to 12 weeks
  Change in delayed matching to sample will be assessed by computerized test using CANTAB (www.cambridgecognition.com).
Change from baseline rapid visual information processing at 12 weeks | 0 to 12 weeks
  Change in rapid visual information processing will be assessed by computerized test using CANTAB (www.cambridgecognition.com).
Adherence to diet supplementation by weekly package return count | 0 to 12 weeks
  Adherence to diet supplementation will be assessed by counts of opened and unopened supplement packets returned each week.

CONTACTS AND LOCATIONS:
Overall Officials: William Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller MG, Hamilton DA, Joseph JA, Shukitt-Hale B. Dietary blueberry improves cognition among older adults in a randomized, double-blind, placebo-controlled trial. Eur J Nutr. 2018 Apr;57(3):1169-1180. doi: 10.1007/s00394-017-1400-8. Epub 2017 Mar 10. PMID 28283823
- [Background] Michalska A, Lysiak G. Bioactive Compounds of Blueberries: Post-Harvest Factors Influencing the Nutritional Value of Products. Int J Mol Sci. 2015 Aug 10;16(8):18642-63. doi: 10.3390/ijms160818642. PMID 26266408
- [Background] Whyte AR, Cheng N, Fromentin E, Williams CM. A Randomized, Double-Blinded, Placebo-Controlled Study to Compare the Safety and Efficacy of Low Dose Enhanced Wild Blueberry Powder and Wild Blueberry Extract (ThinkBlue) in Maintenance of Episodic and Working Memory in Older Adults. Nutrients. 2018 May 23;10(6):660. doi: 10.3390/nu10060660. PMID 29882843
- [Background] Johnson SA, Figueroa A, Navaei N, Wong A, Kalfon R, Ormsbee LT, Feresin RG, Elam ML, Hooshmand S, Payton ME, Arjmandi BH. Daily blueberry consumption improves blood pressure and arterial stiffness in postmenopausal women with pre- and stage 1-hypertension: a randomized, double-blind, placebo-controlled clinical trial. J Acad Nutr Diet. 2015 Mar;115(3):369-377. doi: 10.1016/j.jand.2014.11.001. Epub 2015 Jan 8. PMID 25578927
- [Background] Reis JF, Monteiro VV, de Souza Gomes R, do Carmo MM, da Costa GV, Ribera PC, Monteiro MC. Action mechanism and cardiovascular effect of anthocyanins: a systematic review of animal and human studies. J Transl Med. 2016 Nov 15;14(1):315. doi: 10.1186/s12967-016-1076-5. PMID 27846846
- See also: Duke University School of Medicine — http://medschool.duke.edu/
- See also: U.S. Highbush Blueberry Council — http://www.blueberrycouncil.org